CLINICAL TRIAL: NCT02804126
Title: Effectiveness of Transversus Abdominis Plane Block Versus Quadratus Lumborum Technique in Patients After Cesarean Section
Brief Title: Comparison of Two Pain-treatment Techniques After Cesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michał Borys (Other)
Responsible Party: Sponsor-Investigator, Michał Borys, associate professor, Medical University of Lublin
Organization: Medical University of Lublin (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/85/2016
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cesarean Section; Pain Management; Neuropathic Pain
Keywords: acute pain; transversus abdominis plane block; quadratus lumborum block; neuropathic pain
MeSH Terms: conditions — Agnosia; Neuralgia; Acute Pain | interventions — Bupivacaine; Needles; Acetaminophen; Dipyrone; Ketoprofen; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP (transversus abdominis plane) (Experimental): Ultrasound-guided transversus abdominis plane block at the end of cesarean section
  Interventions: Procedure: TAP (transversus abdominis plane block); Drug: Bupivacaine; Device: Needle; Drug: Paracetamol; Drug: Metamizol; Drug: Ketoprofen; Drug: Morphine
- QL (quadratus lumborum) (Experimental): Ultrasound-guided quadratus lumborum block at the end of cesarean section
  Interventions: Procedure: QL (quadratus lumborum block); Drug: Bupivacaine; Device: Needle; Drug: Paracetamol; Drug: Metamizol; Drug: Ketoprofen; Drug: Morphine

INTERVENTIONS:
Procedure: TAP (transversus abdominis plane block) — ultrasound-guided regional block between abdominal wall muscles to treat acute postoperative pain. Stimuplex Ultra 360 needle will be used and 0.25% bupivacaine administered (0.2 mL/kg).
  Arms: TAP (transversus abdominis plane)
Procedure: QL (quadratus lumborum block) — ultrasound-guided regional block between abdominal wall muscles to treat acute pain, similar to transversus abdominis plane block, but with distribution of local anesthetic towards paravertebral space. Stimuplex Ultra 360 needle will be used and 0.25% bupivacaine administered (0.2 mL/kg).
  Arms: QL (quadratus lumborum)
Drug: Bupivacaine — In both groups (TAP&QL) 0.25% bupivacaine will be given (0.2 mL/kg)
Device: Needle — Ultrasound-guided, Stimuplex ultra 360 needle will be used in the study
Drug: Paracetamol — Intravenous paracetamol will be used (1.0 gram), up to 4 grams per day
Drug: Metamizol — Intravenous metamizol will be used (1.0 gram), up to 4 grams per day
Drug: Ketoprofen — Intravenous ketoprofen will be used (0.1 gram), up to 200 milligrams per day
Drug: Morphine — Intravenous morphine (5 mg) will be given when pain exceeds 40 mm in VAS (maximum 2 doses per day)

SUMMARY:
Comparison of two types of analgesia after cesarean section.

All patients will anaesthetised with spinal technique. Ultrasound-guided transversus abdominis plane or quadratus lumborum block to treat postoperative pain. Postoperative pain will measured with visual-analogue scale (VAS). 1, 2, 6 months after surgery each patient will be called to assess neuropathic pain with Neuropathic Pain Symptom Inventory (NPSI).

DETAILED DESCRIPTION:
Written consent will be obtained before the cesarean section. Only subarachnoidally anaesthetised patients may participate in the study. Pencil-point spinal needle and bupivacaine (Marcaine Heavy Spinal 0.5 %) will be used.

At the end of surgery ultrasound-guided regional block will be performed. Each patient will be randomly allocated to one of the treated group: transversus abdominis plane block (TAP) or quadratus lumborum (QL). Patients receive 0.2 mL of local anesthetic solution (0.25 % bupivacaine) on each side.

Postoperative pain will be measured with VAS (visual-analogue scale) 2, 4, 8, 12 and 24 hours after the end of operation.

Paracetamol, metamizol, ketoprofen may be given as required. Whenever pain exceeds 40 (VAS) 5 mg of morphine will be given intravenously (maximum two dosages per day).

1, 3, 6 months patients will be called to assess neuropathic pain. Neuropathic Pain Symptom Inventory (NPSI) will be used.

ELIGIBILITY:
Inclusion Criteria:

* obtained consent
* singleton pregnancy
* subarachnoid anaesthesia

Exclusion Criteria:

* coagulopathy
* allergy to to local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain measured with VAS | up to 24 hours after surgery
  Acute pain measured with VAS (visual-analogue scale).

SECONDARY OUTCOMES:
Neuropathic pain assessed with NPSI | 6 months from the surgery
  Neuropathic pain occurrence with Neuropathic Pain Symptom Inventory (NPSI)

CONTACTS AND LOCATIONS:
Overall Officials: Miroslaw Czuczwar, MD, PhD, Study Chair — II Department of Anesthesiology and Intensive Care Medial University of Lublin
Locations (1):
- II Department of Anesthesia and Intensive Care, Lublin, Poland

REFERENCES:
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Kadam VR. Ultrasound guided quadratus lumborum block or posterior transversus abdominis plane block catheter infusion as a postoperative analgesic technique for abdominal surgery. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):130-1. doi: 10.4103/0970-9185.150575. No abstract available. PMID 25788791
- [Background] Kanazi GE, Aouad MT, Abdallah FW, Khatib MI, Adham AM, Harfoush DW, Siddik-Sayyid SM. The analgesic efficacy of subarachnoid morphine in comparison with ultrasound-guided transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2010 Aug;111(2):475-81. doi: 10.1213/ANE.0b013e3181e30b9f. Epub 2010 May 20. PMID 20488929